CLINICAL TRIAL: NCT06434285
Title: Development of a 4Pi Framework-based Questionnaire to Evaluate Service User and Carer Involvement Experience in SLaM
Brief Title: A 4Pi Questionnaire for Service User and Carer Involvement Experience
Acronym: 4PiQ
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 321452
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire development — Cognitive interviewing group will be run to inform questionnaire development.

SUMMARY:
Service user (SU) and carer involvement in planning healthcare services and improving their quality is crucial and required by the NHS. Research has shown that SUs and carers can greatly benefit healthcare; however, effective involvement can be challenging due to barriers such as language, lack of training or support, and undervaluing the input of patients and the public compared to that of professionals.

The 4Pi framework sets out standards for good involvement practices by focusing on principles such as respect and inclusivity, shared purposes, diversity, accurate planning, and ensuring involvement leads to improvements in people's lives.

This study, funded by King's Health Partners, aims to take the 4Pi framework a step further by developing a questionnaire to evaluate how well patients and carers are involved in improving mental health services. The researchers will work closely with SUs and carers to create this questionnaire, with the ultimate goal to ensure that involvement in healthcare leads to real, positive changes for everyone involved.

The research questions for the study is: to what extent, from SUs and carers' perspectives, is the questionnaire understandable and successful in capturing the meaning of 4Pi domains?

To be eligible for the study, participants need to be at least 18 years old and have experience of involvement activities/projects in SLaM. Researchers, SUs, and carers will define the questionnaire to ensure it is understandable, comprehensive, and feasible; this will be done via virtual (or in person at Denmark Hill/King's College London campus depending on participants' preferences) group interviews. The questionnaire will then be piloted on a small sample of individuals, and the final questionnaire refined based on any potential additional feedback from them.

This study is part of the King's Improvement Science programme's research portfolio that is funded by King's Health Partners.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years old;
2. have experience of being involved in service involvement activities in SLaM NHS Foundation Trust.

Exclusion Criteria:

a) No experience of being involved in service improvement activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Service users and carers with experience in service involvement activities.
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2024-06-24 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | Day 1